CLINICAL TRIAL: NCT04131387
Title: The Safety and Efficacy of Micro-energy Ultrasound Therapy in the Treatment of Female Stress Urinary Incontinence: A Multi-center Randomized Clinical Trial
Brief Title: The Safety and Efficacy of Micro-energy Ultrasound Therapy in the Treatment of Female Stress Urinary Incontinence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-341
Record Dates: First submitted 2019-10-14; First posted 2019-10-18 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2019-10

CONDITIONS: Female Stress Urinary Incontinence
Keywords: Female Stress Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): After installing the disposable treatment head coat, the pelvic floor muscles, ligaments, etc. were treated with an ultrasonic therapeutic apparatus; after the treatment, the disposable treatment head coat was removed. Treated twice a week for 6 weeks.
  Interventions: Device: LIPUS-1
- Control Group (Placebo Comparator): The placebo was treated with an ultrasound therapy device and used in the same manner as the test group.
  Interventions: Device: LIPUS-2

INTERVENTIONS:
Device: LIPUS-1 — After installing the disposable treatment head coat, the pelvic floor muscles, ligaments, etc. were treated with an ultrasonic therapeutic apparatus; after the treatment, the disposable treatment head coat was removed. Treated twice a week for 6 weeks.
  Arms: Test Group
Device: LIPUS-2 — The placebo was treated with an ultrasound therapy device and used in the same manner as the test group.
  Arms: Control Group

SUMMARY:
The Safety and Efficacy of Micro-energy Ultrasound Therapy in the Treatment of Female Stress Urinary Incontinence: A Multi-center Randomized Trail

DETAILED DESCRIPTION:
1. Study purpose: To evaluate the safety and efficacy of micro-energy ultrasound therapy in the treatment of female stress urinary incontinence
2. Study design: This is a randomized, double-blind, controlled, multi-center clinical trial
3. Study subjects: Females with mild to moderate stress urinary incontinence
4. Number of subjects: 60
5. Study center: The Second Affiliated Hospital, School of Medicine, Zhejiang University
6. Treatment methods:

Test group: After installing the disposable treatment head coat, the pelvic floor muscles, ligaments, etc. were treated with an ultrasonic therapeutic apparatus; after the treatment, the disposable treatment head coat was removed. Patients were treated twice a week for 6 weeks.

Control group: The placebo was treated with an ultrasound therapy device and used in the same manner as the test group.

ELIGIBILITY:
Inclusion Criteria:

1. patients diagnosed as mild to moderate female stress urinary incontinence in our hospital;
2. other conservative treatments are ineffective or have poor results, and the operator is not considered for the time being;
3. volunteer to participate in this clinical trial, complied with the requirements of this study and signed the informed consent form.

Exclusion Criteria:

1. other types of urinary incontinence;
2. blood routines indicate acute and chronic blood system diseases;
3. B-ultrasound suggests other gynecological diseases;
4. combine uncontrollable diseases such as diabetes, hypertension, and cardiovascular diseases;
5. previous or current history of pelvic surgery and radiotherapy and chemotherapy;
6. the investigator determined that it is not suitable for this clinical trial.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
The score of ICI-Q-SF | change from baseline level at 2 months after treatment
  measure the international committee of incontinence brief list of urinary incontinence by a questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China